CLINICAL TRIAL: NCT04453319
Title: Efficacy of Negative Pressure Wound Closure Therapy by PICO System in Prevention of Complications of Femoral Artery Exposure
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Mansoura University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: RP.19.12.52.R1 - 2020/01/31
Record Dates: First submitted 2020-06-21; First posted 2020-07-01 (Actual); Last update posted 2020-07-01 (Actual); Status verified 2020-06

CONDITIONS: Wound Infection; Wound Surgical
MeSH Terms: conditions — Wound Infection; Surgical Wound | interventions — Bandages

STUDY DESIGN:
Intervention Model Description: Randomized Comparative study
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Block randomization
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Application of the device (PICO) (Experimental): PICO® is a disposable, single-use pump without a canister that generates an effective, non-adjustable, negative pressure of -80 mmHg and that can be used for up to 7 days.(-1113) It incorporates leak detection and low battery indicators and is connected to a 4-layer absorbent dressing that primarily removes wound exudates through evaporative loss. The mechanism of action has been postulated to occur because of the combined effects of a reduction in the frequency of dressing changes, a reduction in stress concentration in the tissue surrounding the incision, and an enhancement in the appositional strength of the incision line, thus reducing dead space and minimizing the risk of wound contamination.(14) PICO® has also been demonstrated to enhance lymphatic clearance and decrease the risk of hematomas or seromas
  Interventions: Procedure: Femoral Wound Closure and dressing
- Conventional Dressing of the femoral wound (No Intervention): Conventional Dressing of the femoral wound

INTERVENTIONS:
Procedure: Femoral Wound Closure and dressing — Femoral Wound Closure and dressing
  Arms: Application of the device (PICO)

SUMMARY:
Evaluate negative pressure wound closure therapy by PICO system in Prevention of complications of femoral artery exposure.

DETAILED DESCRIPTION:
INTRODUCTION:

Wound infection is a very common complication in patients who undergo femoral artery exposure. It can lead to prolonged hospital stays, increased healthcare expenditures, admission times, graft failure, and limb loss and is recognized as a significant cause of postoperative morbidity and mortality.

Negative pressure wound therapy (NPWT) has been developped as a method for reducing the risk of wound complications and is the wound dressing of choice in many vascular procedures during the arterial exposure.

The idea of NPWT is a therapeutic technique wherein subatmospheric pressure is applied to a wound using a sealed wound dressing that is connected to a vacuum pump, which can be continuously or intermittently applied.

The mechanism of NPWT, is that it facilitates wound healing by decreasing the bacterial burden; promoting granulation tissue formation, capillary blood flow, endothelial proliferation, and angiogenesis; and restoring the integrity of the capillary basement membrane.

The clinical efficacy of NPWT for closed incisions has been extensively studied in surgical disciplines such as orthopedics, cardiothoracic, and plastic surgery, and its use in promoting wound healing and improving patient outcomes has been validated. The use of vacuum-assisted closure dressings (PICO system) is currently no evidenced that supports the use PICO system of for lower limb femoral incisions. Therefore, we aimed to evaluate the outcomes of PICO system in preventing wound complication in patients with femoral artery exposure.

Aim of the work Evaluate negative pressure wound closure therapy by PICO system in Prevention of complications of femoral artery exposure.

Outcome

Primary outcomes:

Infection Hematoma seroma

Secondary outcomes:

Wound Dehiscence. Patients and methods Study location: The study will be conducted at the department of vascular surgery in Mansoura university hospitals Type of study: Randomized controlled Prospective study Study duration: 2 years: 2019-2021 Sample size: 250 patients n=(Z^2 p(1-p))/d^2 Where: Z= 1.96 at 95% confidence level, P= expected prevalence, d= precision (margin of error)

Study population: The study will be conducted in all patients suspected to femoral artery exposure whatever the type of surgery Inclusion criteria: all patients suspected to femoral artery exposure whatever the type of surgery Exclusion criteria who can't give consent (unconscious)? Those with mental or behavioral disorders will be excluded. Consent: Patients after signing informed consent that possible complication from the procedure ought to happen and what are the alternatives.

Data collection: The demographics, Symptoms and preoperative clinical data will be collected History Data: included patient's demographics, underlying medical conditions, any previous associated morbidity.

Examination: Arterial assessments. Laboratory: Blood picture, Blood sugar level, Kidney functions, Liver functions and Coagulation profile.

Imaging: Duplex US and CTA Method of Randomization: Block randomization: Two elements A for Application of the device, B for conventional dressing A A B B A B A B A B B A B B A A B A B A B A A B Technique After closure of Femoral wound the PICO system is applied for up to 5-7 days. PICO® is a disposable, single-use pump without a canister that generates an effective, non-adjustable, negative pressure of -80 mmHg and that can be used for up to 7 days.(-1113) It incorporates leak detection and low battery indicators and is connected to a 4-layer absorbent dressing that primarily removes wound exudates through evaporative loss. The mechanism of action has been postulated to occur because of the combined effects of a reduction in the frequency of dressing changes, a reduction in stress concentration in the tissue surrounding the incision, and an enhancement in the appositional strength of the incision line, thus reducing dead space and minimizing the risk of wound contamination.(14) PICO® has also been demonstrated to enhance lymphatic clearance and decrease the risk of hematomas or seromas(15) Follow up Every patient will be followed every week till first month, then every 3 months till 1 years.

Hemodynamic improvement was assessed by ankle brachial pressure index (ABI), performed before and after the procedure and every 3 months.

Evaluation made to determine wound complications (Infection, Hematoma, seroma and wound dehiscence)

Statistical analysis The data will be analyzed using Statistical Package for the Social Sciences. The numerical outcomes e.g. age is calculated as mean. Gender will be recorded as frequency and percentage. Chi Square test is applied to assess the association of various parameters. The results will be considered statistically significant if the p-value is found to be less than or equal to 0.05.

ELIGIBILITY:
Inclusion Criteria:

* All femoral artery exposure whatever the type of surgery

Exclusion Criteria:

* who can't give consent (unconscious)
* Those with mental or behavioral disorders

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 250 (Estimated)
Dates: Start 2020-01-31 (Actual); Primary Completion 2021-01-30 (Estimated); Study Completion 2021-01-30 (Estimated)

PRIMARY OUTCOMES:
Infection | 12 months
  Clinical( fever, collection) and Radiological
Hematoma | 12 months
  Blood collected under the suture line
seroma | 12 months
  Fluid collected under the suture line

SECONDARY OUTCOMES:
Wound Dehiscence | 12 Months
  a wound ruptures along a surgical incision

CONTACTS AND LOCATIONS:
Locations (1):
- Mansoura, Al Mansurah, Mansoura University, Egypt

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Correia RM, Nakano LC, Vasconcelos V, Cristino MA, Flumignan RL. Prevention of infection in peripheral arterial reconstruction of the lower limb. Cochrane Database Syst Rev. 2025 Oct 29;10(10):CD015022. doi: 10.1002/14651858.CD015022.pub2. PMID 41159585